CLINICAL TRIAL: NCT00442715
Title: Exercise Challenge Test in 3-6 Years Old Asthmatic Children
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4400-YY-CTIL
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2007-03-06 (Estimated); Status verified 2007-03

CONDITIONS: Asthma
Keywords: Exercise-induced asthma,; early childhood;; spirometry,; exercise challenge; Data from preschool children who were referred to the Pediatric; Pulmonary Clinic over a 1-year period were recruited
MeSH Terms: conditions — Asthma; Asthma, Exercise-Induced

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Exercise chalenge test

SUMMARY:
Vigorous exercise is known to cause transient bronchoconstriction in school children with asthma, many of whom initially have normal lung function at rest. The presence and extent of this phenomena in early childhood is difficult to recognize, because exercise induced bronchoconstriction (EIB) may not limit the child's performance and the child may fail to notice the symptoms until taking part in organized or competitive sport. Conversely, as children do participate in vigorous activities all day long, severe EIB may provoke a crucial disabling condition in the child.

In school children the exercise challenge test (ECT) is a well standardized test and is used to make a diagnosis of asthma because it is able to discriminate between asthma and other chronic breathing illnesses of childhood and is also used to determine the effectiveness and optimal dosages of medications prescribed to prevent EIB.

The test includes is a controlled run on a motor-driven treadmill followed by scheduled multiple spirometry maneuvers. This procedure was never been tested and may not be suitable for the preschool age.

In this study we assumed that a free-run test which combined with measurements of duplicate spirometry-sets would be the most convenient way to test young children.

The aims of this study are a) to examine the feasibility of a free-run protocol (according to the ATS/ERS recomendations), followed by duplicate spirometry measurements in early childhood.

b) to explore the existence of exercise induced bronchoconstriction in young children (age 3-6 years old) with respiratory symptoms.

DETAILED DESCRIPTION:
Method:

The children are to come in comfortable clothes and running shoes, having consumed no more than a light meal and having had pulmonary medications withdrawn as described above. A parent, a pediatric pulmonary physician and a technician is present throughout the test. Each child undergoes a physical examination to exclude evidence of wheeze, and baseline spirometry was performed. The children are asked to run freely back and forth (without a nose-clip) in a 50m long corridor next to the pulmonary laboratory. The target is to achieve 6 minutes of "free run" to increase hart-rate to 80% in the maximum for at least 4 minutes according to ATS/ERS recommendations for exercise challenge test in older children [1]. An adult (parent/technician/ physician) will run with the child to encourage him/her to continue running. Heart-rate and O2-saturation is monitored continuously throughout the run using a portable mobile pulse-oximeter monitor (Nonin medical, INC, model 2500, Minneapolis, USA).

Spirometry is measured according to the recommendations for preschool children [2], with a commercial ZAN100 Spirometer situated in the pediatric pulmonary laboratory, by a skilled technician. Measurements are performed in the standing position, without nose-clip (for comfort of the child) until two consecutive technically acceptable curves are achieved. After the free-run, spiroetmry is measured in duplicate sets at 1, 3, 5, 10 and 20 minutes post-exercise [1]. The better of the two curves is selected as the representative value at each interval, but differences between the two values of FEV1 has to be <5%. The following signs are monitored by the pulmonologist: wheeze and prolonged expiration on auscultation over the trachea and two zones of both lungs (upper front and lower back). Cough, shortness of breath, or perceived breathlessness within 20 minutes after the run were noted.

Analysis: Technically acceptable spirometry maneuvers are analyzed. Baseline values are first compared to the spirometry values with relation to height derived from the indices in 109 healthy children in our previous study [3].

Following exercise, best spirometry values for each interval are compared to baseline values. Exercise response was defined as the greatest decrease in FEV1 expressed as a percentage of the baseline values. A bronchoconstriction response to exercise is considered as positive when the FEV1 decrease from baseline was greater than 13% [4]. Student's paired t-test is used for comparison of data between each spirometry index and the calculated values for healthy children. A value of p<0.05 was considered significant.

References:

1. Guidelines for Methacholine and Exercise Challenge Testing 1999. The official statements of the American Thoracic Society, adopted by the ATS board of directors, 1999. Am J Respir Crit. Care Med 2000;161:309-329.
2. Aurora P, Stocks J, Oliver C, Saunders C, Castle R, Chaziparasidis G, Bush A; London Cystic Fibrosis Collaboration. Quality control for spirometry in preschool children with and without lung disease. Am J Respir Crit Care Med 2004; 169:1152-1159.
3. Vilozni D, Barak A, Efrati O, Augarten A, Springer C, Yahav Y, Bentur L. The role of computer games in measuring spirometry in healthy and "asthmatic" preschool children. Chest. 2005; 128:1146-115.
4. Godfrey S, Springer C, Bar-Yishay E, Avital A. Cut-off points defining normal and asthmatic bronchial reactivity to exercise and inhalation challenges in children and young adults. Eur Respir J. 1999; 14:659-66.

ELIGIBILITY:
Inclusion Criteria:

* 3.0-6.9 year-old children referred for exercise challenge test by pediatric physicians.

Exclusion Criteria:

* presence of other chronic respiratory conditions (e.g. cystic fibrosis, bronchopulmonary dysplasia); oral or inhaled steroids taken during the previous week; bronchodilator taken within 24 hours prior to the test; wheezing at physical examination prior to exercise test, and baseline FEV1< 70 % predicted.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2006-10; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Daphna Vilozni, PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Pediatric pulmonary unit, The Edmod and Lili Safra children's Hospital, Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Vilozni D, Barak A, Efrati O, Augarten A, Springer C, Yahav Y, Bentur L. The role of computer games in measuring spirometry in healthy and "asthmatic" preschool children. Chest. 2005 Sep;128(3):1146-55. doi: 10.1378/chest.128.3.1146. PMID 16162700
- [Background] Aurora P, Stocks J, Oliver C, Saunders C, Castle R, Chaziparasidis G, Bush A; London Cystic Fibrosis Collaboration. Quality control for spirometry in preschool children with and without lung disease. Am J Respir Crit Care Med. 2004 May 15;169(10):1152-9. doi: 10.1164/rccm.200310-1453OC. Epub 2004 Mar 17. PMID 15028561
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836
- [Background] Godfrey S, Springer C, Bar-Yishay E, Avital A. Cut-off points defining normal and asthmatic bronchial reactivity to exercise and inhalation challenges in children and young adults. Eur Respir J. 1999 Sep;14(3):659-68. doi: 10.1034/j.1399-3003.1999.14c28.x. PMID 10543290